CLINICAL TRIAL: NCT02958956
Title: Cohort Study of Pioglitazone and Cancer Incidence in Patients With Diabetes Mellitus
Brief Title: Cohort Study of Pioglitazone and Cancer Incidence in Participants With Diabetes Mellitus.
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: AD-4833_403A; EUPAS10335 (Registry Identifier: EU PAS)
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus, Type 2, Cancer
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ever User of Pioglitazone: Ever user of pioglitazone was defined as having filled 2 prescriptions for the drug within a 6-month period.
  Interventions: Drug: Pioglitazone
- Never User of Pioglitazone: Never user of pioglitazone, which included participants receiving no diabetes medications, with fewer than 2 pioglitazone prescription fills in a 6-month period, and with use of diabetes medications other than pioglitazone.

INTERVENTIONS:
Drug: Pioglitazone — Participants with diabetes who were members of the KPNC registry, and had received at least 2 prescriptions for pioglitazone within a 6-month period were followed up to 15.5 years (1997-2012) in this observational study 1.
  Groups: Ever User of Pioglitazone

SUMMARY:
The purpose of this study was to evaluate whether treatment with pioglitazone is associated with risk of incident cancer at the 10 most common sites in a cohort of participants with recognized diabetes.

DETAILED DESCRIPTION:
The study enroll a large population of approximately 252467 participants. The study would analyze association of cancer and pioglitazone in 2 cohorts based on the usage of pioglitazone. Participants in were originally planned to be followed-up from January 1, 1997 to December 31, 2005. Based on the discussion with advisory board, it was recommended to increase the study population and duration of follow-up. The follow-up period was extended to June 30, 2012 for the study.

This multi-center trial was conducted in the United States of America. The overall time to participate in this study was approximately 15.5 years. Participants were followed-up from January 1, 1997 up to June 30, 2012 for the assessment of cancer risk associated with pioglitazone use.

ELIGIBILITY:
Inclusion Criteria:

1. has been in the KPNC diabetes registry Diabetes Mellitus (DM) registry, aged 40 years or older and are members of KPNC as of January 1, 1997, or
2. has been in the DM registry, reached aged 40 years between January 1, 1997 and June 30, 2005 and are KPNC members on their 40th birthday, or
3. has joined KPNC after January 1, 1997, aged 40 years or older when they are identified by the DM registry between January 1, 1997 and June 30, 2005.

Exclusion Criteria: 1. Age less than (<) 40 years during study period. 2. No KPNC medication benefits at the time of entry into the cohort (baseline) or gap in medication benefit greater than equal to (>=) 4 months that started in the first 4 months after entering in the cohort.

3. Gap in KPNC membership >= 4 months that started in the first 4 months after entering in the cohort.

4. Participant with a diagnosis of Human immunodeficiency virus (HIV). 5. Participants with evidence of selected surgeries for some cancer sites. 6. All prevalent cancers at baseline, that is, all participants ever diagnosed with cancer other than non-melanoma skin cancer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a historical diagnosis of Type 2 diabetes mellitus (T2DM) with pioglitazone exposure identified from the Kaiser Permanente of Northern California(KPNC) Diabetes Registry (with or without diabetes) and had completed Member Health Survey (MHS) were enrolled in the epidemiology study.
Sampling Method: Probability Sample
Enrollment: 236507 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2015-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- See also: Interim Results Report — https://www.takeda.com/siteassets/en-us/home/external-reference/clinicaltrials.gov/ad-4833-403-fum_35.4_kpnc_interim_results_report-2011-12-07.pdf
- See also: 10 yr Study Report — https://www.takeda.com/siteassets/en-us/home/external-reference/clinicaltrials.gov/ad4833-403_kpnc_10_common_cancers_10-yr_study_report.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 01 July 1997 to 30 June 2012.
Pre-assignment Details: Participants with a historical diagnosis of T2DM with pioglitazone exposure identified from the Kaiser Permanente of Northern California(KPNC) Diabetes Registry were enrolled in this observational study.
Period: Overall Study
Arm/Group | Ever User of Pioglitazone | Never User of Pioglitazone
Started | 38190 | 198317
Completed | 38190 | 198317
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population consisted of Type 2 diabetes mellitus (T2DM) participants who were identified from the Kaiser Diabetes Registry, were included in the membership database, medication benefit database, hospitalization and surgery procedures databases, cancer registry database merged along with data in the diabetes registry were evaluable for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ever User of Pioglitazone | Never User of Pioglitazone | Total
Number analyzed (Participants) | 38190 | 198317 | 236507
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (10.4) | 59.7 (12.2) | 59.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17632 | 92552 | 110184
  Male | 20558 | 105765 | 126323
Race/Ethnicity, Customized [Number; unit: Participants]
  Non-Hispanic white | 18717 | 99641 | 118358
  African American | 3667 | 19931 | 23598
  Asian or Pacific Islander | 5695 | 26637 | 32332
  Hispanic | 5144 | 21554 | 26698
  Other | 2129 | 10549 | 12678
  Missing | 2838 | 20005 | 22843
Smoking [Number; unit: Participants]
  Current smoking | 7929 | 37401 | 45330
  Missing | 30261 | 160916 | 191177
Income [Number; unit: Participants] — Income was categorized as high and low based on whether the annual household income lied above or below the average census block median income for the cohort (59,000 US Dollars).
  Participants
    Low | 20379 | 107007 | 127386
    High | 17125 | 86384 | 103509
    Missing | 686 | 4926 | 5612
Renal function [Number; unit: Participants] — Renal function was measured based on the levels of creatinine: normal creatinine (less than [<] 1.5 milligram per deciliter [mg/dL] for males and <1.4 mg/dL for females) and elevated creatinine (greater than or equal to [>=] 1.5 mg/dL for males and >=1.4 mg/dL for females).
  Participants
    Normal creatinine | 29476 | 156510 | 185986
    Elevated creatinine | 1495 | 16234 | 17729
    Missing | 7219 | 25573 | 32792
Congestive Heart Failure [Number; unit: Participants]
  Congestive Heart Failure | 1070 | 12602 | 13672
  Missing | 37120 | 185715 | 222835
Baseline Glycosylated Hemoglobin (HbA1c) [Number; unit: Participants]
  <7.0 percent (%) | 6832 | 63867 | 70699
  7.0-7.9% | 6594 | 34579 | 41173
  8.0-8.9% | 4514 | 17971 | 22485
  9.0-9.9% | 3451 | 12342 | 15793
  >=10.0% | 8390 | 29836 | 38226
  Missing | 8409 | 39722 | 48131
Time since diabetes diagnosis [Number; unit: Participants]
  0-4 years | 22835 | 134209 | 157044
  5-9 years | 3148 | 9554 | 12702
  >= 10 years | 2993 | 17300 | 20293
  Missing | 9214 | 37254 | 46468

OUTCOME MEASURES:

1. Primary Outcome: Hazard Ratio of the 10 Most Common Cancers Associated With Ever Use of Pioglitazone
Description: The hazard ratio of the 10 most common cancers: prostate, female breast, lung/bronchus, endometrial, colon, non-Hodgkin lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma associated with ever use of pioglitazone. Cox proportional hazards regression modeling was used to provide point and interval estimates of the relative hazard of the 10 most common cancers associated with ever use of pioglitazone. In all regression analyses, these measures of exposure to pioglitazone were treated as time-dependent covariates and time since entry into the cohort was the time scale.
Time Frame: 15 years 5 months
Population: Analysis population included T2DM participants who were identified from the KPNC Diabetes Registry in the study 1.
Measure: Number (95% Confidence Interval); unit: Ratio
Groups:
- Full Cohort: Participants with diabetes who were members of the KPNC registry, who received (ever use) at least 2 prescriptions for pioglitazone within a 6-month period or who did not receive pioglitazone were followed up to 15.5 years (1997-2012) in this observational study.
Arm/Group | Full Cohort
Number analyzed (Participants) | 236507
Ratio
  Prostate | 1.13 [1.02 to 1.26]
  Breast | 1.00 [0.88 to 1.13]
  Lung/Bronchus | 1.00 [0.87 to 1.15]
  Colon | 0.91 [0.78 to 1.05]
  Non-Hodgkin Lymphoma | 1.00 [0.81 to 1.23]
  Corpus Uteri | 0.88 [0.71 to 1.09]
  Pancreatic | 1.41 [1.16 to 1.71]
  Kidney/Renal Pelvis | 0.95 [0.76 to 1.18]
  Rectum | 0.81 [0.60 to 1.08]
  Melanoma | 1.15 [0.91 to 1.46]

2. Primary Outcome: Number of 10 Most Common Cancers Associated Cases
Description: Number of 10 most common cancer cases are reported in this measure: prostate, female breast, lung/bronchus, endometrial, colon, non-Hodgkin lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma.
Time Frame: 15 years 5 months
Population: Analysis population included T2DM participants who were identified from the KPNC Diabetes Registry in the study 1.
Measure: Number; unit: Cases
Arm/Group | Ever User of Pioglitazone | Never User of Pioglitazone
Number analyzed (Participants) | 38190 | 198317
Cases
  Prostate | 476 | 3307
  Breast | 320 | 2478
  Lung/Bronchus | 282 | 2300
  Colon | 233 | 1844
  Non-Hodgkin Lymphoma | 120 | 839
  Corpus Uteri | 118 | 799
  Pancreatic | 164 | 648
  Kidney/Renal Pelvis | 110 | 690
  Rectum | 59 | 570
  Melanoma | 102 | 594

3. Secondary Outcome: Hazard Ratio of the 10 Most Common Cancers Associated With Time Since First Use of Pioglitazone
Description: The hazard ratio of the 10 most common cancers: prostate, female breast, lung/bronchus, endometrial, colon, non-Hodgkin lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma associated with time since first use of pioglitazone. The various times since initiation include <12 months ago, 12-23 months ago, 24-35 months ago, 36-47 months ago, 48-83 months ago and 84+ months ago. Cox proportional hazards regression modeling was used to provide point and interval estimates of the time since first use. In all regression analyses, these measures of exposure to pioglitazone were treated as time-dependent covariates and time since entry into the cohort was the time scale.
Time Frame: 15 years 5 months
Population: Analysis population included T2DM participants who were identified from the KPNC Diabetes Registry in the study 1.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Full Cohort
Number analyzed (Participants) | 236507
Ratio
  Prostate: <12 months ago | 0.92 [0.73 to 1.17]
  Prostate: 12-23 months ago | 1.18 [0.94 to 1.47]
  Prostate: 24-35 months ago | 1.21 [0.96 to 1.52]
  Prostate: 36-47 months ago | 1.36 [1.07 to 1.71]
  Prostate: 48-83 months ago | 1.04 [0.86 to 1.26]
  Prostate: 84+ months ago | 1.23 [0.95 to 1.59]
  Breast: <12 months ago | 1.00 [0.76 to 1.31]
  Breast: 12-23 months ago | 0.84 [0.62 to 1.14]
  Breast: 24-35 months ago | 1.04 [0.77 to 1.39]
  Breast: 36-47 months ago | 0.77 [0.54 to 1.10]
  Breast: 48-83 months ago | 1.03 [0.83 to 1.28]
  Breast: 84+ months ago | 1.38 [1.06 to 1.80]
  Lung/Bronchus: <12 months ago | 0.82 [0.59 to 1.14]
  Lung/Bronchus: 12-23 months ago | 1.12 [0.84 to 1.50]
  Lung/Bronchus: 24-35 months ago | 1.13 [0.84 to 1.53]
  Lung/Bronchus: 36-47 months ago | 1.04 [0.75 to 1.45]
  Lung/Bronchus: 48-83 months ago | 0.95 [0.74 to 1.20]
  Lung/Bronchus: 84+ months ago | 0.96 [0.70 to 1.31]
  Colon: <12 months ago | 0.62 [0.41 to 0.92]
  Colon: 12-23 months ago | 0.79 [0.55 to 1.14]
  Colon: 24-35 months ago | 1.35 [1.00 to 1.81]
  Colon: 36-47 months ago | 0.81 [0.55 to 1.19]
  Colon: 48-83 months ago | 0.97 [0.76 to 1.24]
  Colon: 84+ months ago | 0.79 [0.56 to 1.12]
  Non-Hodgkin Lymphoma: <12 months ago | 1.15 [0.75 to 1.76]
  Non-Hodgkin Lymphoma: 12-23 months ago | 1.44 [0.97 to 2.14]
  Non-Hodgkin Lymphoma: 24-35 months ago | 0.92 [0.56 to 1.53]
  Non-Hodgkin Lymphoma: 36-47 months ago | 0.79 [0.44 to 1.40]
  Non-Hodgkin Lymphoma: 48-83 months ago | 0.70 [0.46 to 1.06]
  Non-Hodgkin Lymphoma: 84+ months ago | 0.98 [0.61 to 1.56]
  Corpus Uteri: <12 months ago | 0.91 [0.58 to 1.43]
  Corpus Uteri: 12-23 months ago | 0.97 [0.62 to 1.53]
  Corpus Uteri: 24-35 months ago | 0.65 [0.37 to 1.16]
  Corpus Uteri: 36-47 months ago | 0.90 [0.54 to 1.52]
  Corpus Uteri: 48-83 months ago | 0.99 [0.70 to 1.41]
  Corpus Uteri: 84+ months ago | 0.94 [0.59 to 1.51]
  Pancreatic: <12 months ago | 2.27 [1.61 to 3.20]
  Pancreatic: 12-23 months ago | 1.31 [0.85 to 2.01]
  Pancreatic: 24-35 months ago | 1.13 [0.71 to 1.82]
  Pancreatic: 36-47 months ago | 1.28 [0.80 to 2.04]
  Pancreatic: 48-83 months ago | 1.14 [0.82 to 1.60]
  Pancreatic: 84+ months ago | 1.39 [0.93 to 2.07]
  Kidney/Renal Pelvis: <12 months ago | 0.75 [0.43 to 1.30]
  Kidney/Renal Pelvis: 12-23 months ago | 0.59 [0.32 to 1.11]
  Kidney/Renal Pelvis: 24-35 months ago | 1.14 [0.71 to 1.83]
  Kidney/Renal Pelvis: 36-47 months ago | 1.16 [0.71 to 1.90]
  Kidney/Renal Pelvis: 48-83 months ago | 1.01 [0.71 to 1.44]
  Kidney/Renal Pelvis: 84+ months ago | 0.90 [0.55 to 1.50]
  Rectum: <12 months ago | 0.67 [0.34 to 1.29]
  Rectum: 12-23 months ago | 0.65 [0.32 to 1.31]
  Rectum: 24-35 months ago | 1.02 [0.56 to 1.86]
  Rectum: 36-47 months ago | 1.27 [0.71 to 2.27]
  Rectum: 48-83 months ago | 0.60 [0.33 to 1.08]
  Rectum: 84+ months ago | 0.87 [0.42 to 1.81]
  Melanoma: <12 months ago | 1.03 [0.60 to 1.76]
  Melanoma: 12-23 months ago | 1.37 [0.85 to 2.21]
  Melanoma: 24-35 months ago | 1.02 [0.57 to 1.83]
  Melanoma: 36-47 months ago | 1.45 [0.87 to 2.40]
  Melanoma: 48-83 months ago | 0.96 [0.62 to 1.47]
  Melanoma: 84+ months ago | 1.47 [0.91 to 2.36]

4. Secondary Outcome: Number of 10 Most Common Cancers Cases by Time Since First Use of Pioglitazone
Description: Number of 10 most common cancer cases: prostate, female breast, lung/bronchus, endometrial, colon, non-Hodgkin lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma associated with time since first use of pioglitazone. Time since initiation of pioglitazone was categorized as <12 months ago, 12-23 months ago, 24-35 months ago, 36-47 months ago, 48-83 months ago and 84+ months ago.
Time Frame: 15 years 5 months
Population: Analysis population included T2DM participants who were identified from the KPNC Diabetes Registry in the study 1. The unexposed arm was not planned to be analyzed for this outcome measure.
Measure: Number; unit: Cases
Arm/Group | Ever User of Pioglitazone
Number analyzed (Participants) | 38190
Cases
  Prostate: <12 months ago | 55
  Prostate: 12-23 months ago | 82
  Prostate: 24-35 months ago | 76
  Prostate: 36-47 months ago | 75
  Prostate: 48-83 months ago | 119
  Prostate: 84+ months ago | 69
  Breast: <12 months ago | 42
  Breast: 12-23 months ago | 42
  Breast: 24-35 months ago | 47
  Breast: 36-47 months ago | 31
  Breast: 48-83 months ago | 91
  Breast: 84+ months ago | 67
  Lung/Bronchus: <12 months ago | 32
  Lung/Bronchus: 12-23 months ago | 48
  Lung/Bronchus: 24-35 months ago | 45
  Lung/Bronchus: 36-47 months ago | 37
  Lung/Bronchus: 48-83 months ago | 75
  Lung/Bronchus: 84+ months ago | 45
  Colon: <12 months ago | 22
  Colon: 12-23 months ago | 30
  Colon: 24-35 months ago | 47
  Colon: 36-47 months ago | 26
  Colon: 48-83 months ago | 71
  Colon: 84+ months ago | 37
  Non-Hodgkin Lymphoma: <12 months ago | 21
  Non-Hodgkin Lymphoma: 12-23 months ago | 26
  Non-Hodgkin Lymphoma: 24-35 months ago | 16
  Non-Hodgkin Lymphoma: 36-47 months ago | 12
  Non-Hodgkin Lymphoma: 48-83 months ago | 24
  Non-Hodgkin Lymphoma: 84+ months ago | 21
  Corpus Uteri: <12 months ago | 14
  Corpus Uteri: 12-23 months ago | 20
  Corpus Uteri: 24-35 months ago | 12
  Corpus Uteri: 36-47 months ago | 15
  Corpus Uteri: 48-83 months ago | 36
  Corpus Uteri: 84+ months ago | 21
  Pancreatic: <12 months ago | 33
  Pancreatic: 12-23 months ago | 22
  Pancreatic: 24-35 months ago | 18
  Pancreatic: 36-47 months ago | 19
  Pancreatic: 48-83 months ago | 41
  Pancreatic: 84+ months ago | 31
  Kidney/Renal Pelvis: <12 months ago | 12
  Kidney/Renal Pelvis: 12-23 months ago | 10
  Kidney/Renal Pelvis: 24-35 months ago | 18
  Kidney/Renal Pelvis: 36-47 months ago | 17
  Kidney/Renal Pelvis: 48-83 months ago | 35
  Kidney/Renal Pelvis: 84+ months ago | 18
  Rectum: <12 months ago | 8
  Rectum: 12-23 months ago | 8
  Rectum: 24-35 months ago | 11
  Rectum: 36-47 months ago | 12
  Rectum: 48-83 months ago | 12
  Rectum: 84+ months ago | 8
  Melanoma: <12 months ago | 10
  Melanoma: 12-23 months ago | 18
  Melanoma: 24-35 months ago | 12
  Melanoma: 36-47 months ago | 16
  Melanoma: 48-83 months ago | 24
  Melanoma: 84+ months ago | 22

5. Secondary Outcome: Hazard Ratio of the 10 Most Common Cancers Associated With Duration of Pioglitazone
Description: The hazard ratio of the 10 most common cancers: prostate, female breast, lung/bronchus, endometrial, colon, non-Hodgkin lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma associated with duration of pioglitazone. The duration of pioglitazone was categorized as <12 months, 12-23 months, 24-35 months, 36-59 months, 60+ months. Cox proportional hazards regression modeling was used to provide point and interval estimates of the cumulative duration. In all regression analyses, these measures of exposure to pioglitazone were treated as time-dependent covariates and time since entry into the cohort was the time scale.
Time Frame: 15 years 5 months
Population: Analysis population included T2DM participants who were identified from the KPNC Diabetes Registry in the study 1.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Full Cohort
Number analyzed (Participants) | 236507
Ratio
  Prostate: <12 months | 1.00 [0.84 to 1.19]
  Prostate: 12-23 months | 1.30 [1.08 to 1.57]
  Prostate: 24-35 months | 1.07 [0.84 to 1.35]
  Prostate: 36-59 months | 1.18 [0.96 to 1.45]
  Prostate: 60+ months | 1.16 [0.90 to 1.50]
  Breast: <12 months | 0.84 [0.69 to 1.03]
  Breast: 12-23 months | 1.07 [0.84 to 1.35]
  Breast: 24-35 months | 1.01 [0.75 to 1.35]
  Breast: 36-59 months | 1.06 [0.82 to 1.38]
  Breast: 60+ months | 1.25 [0.93 to 1.68]
  Lung/Bronchus: <12 months | 0.90 [0.73 to 1.12]
  Lung/Bronchus: 12-23 months | 0.98 [0.75 to 1.27]
  Lung/Bronchus: 24-35 months | 0.96 [0.70 to 1.31]
  Lung/Bronchus: 36-59 months | 1.06 [0.81 to 1.40]
  Lung/Bronchus: 60+ months | 1.12 [0.81 to 1.54]
  Colon: <12 months | 0.86 [0.68 to 1.08]
  Colon: 12-23 months | 0.88 [0.66 to 1.18]
  Colon: 24-35 months | 1.03 [0.75 to 1.42]
  Colon: 36-59 months | 0.66 [0.46 to 0.94]
  Colon: 60+ months | 1.05 [0.76 to 1.46]
  Non-Hodgkin Lymphoma: <12 months | 0.93 [0.66 to 1.29]
  Non-Hodgkin Lymphoma: 12-23 months | 1.25 [0.87 to 1.80]
  Non-Hodgkin Lymphoma: 24-35 months | 1.08 [0.69 to 1.70]
  Non-Hodgkin Lymphoma: 36-59 months | 0.72 [0.44 to 1.18]
  Non-Hodgkin Lymphoma: 60+ months | 0.89 [0.53 to 1.49]
  Corpus Uteri: <12 months | 1.01 [0.75 to 1.35]
  Corpus Uteri: 12-23 months | 0.83 [0.55 to 1.25]
  Corpus Uteri: 24-35 months | 0.97 [0.61 to 1.55]
  Corpus Uteri: 36-59 months | 0.78 [0.49 to 1.24]
  Corpus Uteri: 60+ months | 0.73 [0.42 to 1.29]
  Pancreatic: <12 months | 1.48 [1.12 to 1.95]
  Pancreatic: 12-23 months | 1.19 [0.82 to 1.73]
  Pancreatic: 24-35 months | 1.03 [0.64 to 1.66]
  Pancreatic: 36-59 months | 1.63 [1.15 to 2.31]
  Pancreatic: 60+ months | 1.53 [1.00 to 2.33]
  Kidney/Renal Pelvis: <12 months | 0.92 [0.65 to 1.30]
  Kidney/Renal Pelvis: 12-23 months | 0.81 [0.52 to 1.27]
  Kidney/Renal Pelvis: 24-35 months | 0.96 [0.59 to 1.57]
  Kidney/Renal Pelvis: 36-59 months | 0.99 [0.64 to 1.52]
  Kidney/Renal Pelvis: 60+ months | 1.03 [0.63 to 1.68]
  Rectum: <12 months | 0.87 [0.57 to 1.33]
  Rectum: 12-23 months | 0.78 [0.45 to 1.37]
  Rectum: 24-35 months | 0.80 [0.41 to 1.56]
  Rectum: 36-59 months | 0.58 [0.29 to 1.18]
  Rectum: 60+ months | 0.89 [0.43 to 1.82]
  Melanoma: <12 months | 1.06 [0.73 to 1.54]
  Melanoma: 12-23 months | 1.59 [1.08 to 2.33]
  Melanoma: 24-35 months | 1.06 [0.62 to 1.81]
  Melanoma: 36-59 months | 0.80 [0.46 to 1.37]
  Melanoma: 60+ months | 1.46 [0.91 to 2.35]

6. Secondary Outcome: Number of 10 Most Common Cancer Cases by Duration of Pioglitazone
Description: The 10 most common cancer cases included: prostate, female breast, lung/bronchus, endometrial, colon, non-Hodgkin lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma associated with duration of pioglitazone. The duration of pioglitazone was categorized as <12 months, 12-23 months, 24-35 months, 36-59 months, 60+ months.
Time Frame: 15 years 5 months
Population: as for outcome 4
Measure: Number; unit: Cases
Arm/Group | Ever User of Pioglitazone
Number analyzed (Participants) | 38190
Cases
  Prostate: <12 months | 118
  Prostate: 12-23 months | 121
  Prostate: 24-35 months | 72
  Prostate: 36-59 months | 99
  Prostate: 60+ months | 66
  Breast: <12 months | 88
  Breast: 12-23 months | 75
  Breast: 24-35 months | 47
  Breast: 36-59 months | 61
  Breast: 60+ months | 49
  Lung/Bronchus: <12 months | 83
  Lung/Bronchus: 12-23 months | 60
  Lung/Bronchus: 24-35 months | 41
  Lung/Bronchus: 36-59 months | 56
  Lung/Bronchus: 60+ months | 42
  Colon: <12 months | 72
  Colon: 12-23 months | 48
  Colon: 24-35 months | 40
  Colon: 36-59 months | 33
  Colon: 60+ months | 40
  Non-Hodgkin Lymphoma: <12 months | 35
  Non-Hodgkin Lymphoma: 12-23 months | 32
  Non-Hodgkin Lymphoma: 24-35 months | 20
  Non-Hodgkin Lymphoma: 36-59 months | 17
  Non-Hodgkin Lymphoma: 60+ months | 16
  Corpus Uteri: <12 months | 43
  Corpus Uteri: 12-23 months | 24
  Corpus Uteri: 24-35 months | 19
  Corpus Uteri: 36-59 months | 19
  Corpus Uteri: 60+ months | 13
  Pancreatic: <12 months | 54
  Pancreatic: 12-23 months | 28
  Pancreatic: 24-35 months | 18
  Pancreatic: 36-59 months | 36
  Pancreatic: 60+ months | 25
  Kidney/Renal Pelvis: <12 months | 32
  Kidney/Renal Pelvis: 12-23 months | 20
  Kidney/Renal Pelvis: 24-35 months | 17
  Kidney/Renal Pelvis: 36-59 months | 23
  Kidney/Renal Pelvis: 60+ months | 18
  Rectum: <12 months | 21
  Rectum: 12-23 months | 13
  Rectum: 24-35 months | 9
  Rectum: 36-59 months | 8
  Rectum: 60+ months | 8
  Melanoma: <12 months | 25
  Melanoma: 12-23 months | 29
  Melanoma: 24-35 months | 14
  Melanoma: 36-59 months | 14
  Melanoma: 60+ months | 20

7. Secondary Outcome: Hazard Ratio of the 10 Most Common Cancers Associated With Cumulative Dose of Pioglitazone
Description: The hazard ratio of the 10 most common cancers: prostate, female breast, lung/bronchus, endometrial, colon, non-Hodgkin lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma associated with dose of pioglitazone. The various doses include 1-9000 mg, 9001-25000 mg, 25001-50000 milligram (mg) and greater than or equal to (>=) 50001 mg. Cox proportional hazards regression modeling was used to provide point and interval estimates of the dose. In all regression analyses, these measures of exposure to pioglitazone were treated as time-dependent covariates and time since entry into the cohort was the time scale.
Time Frame: 15 years 5 months
Population: Analysis population included T2DM participants who were identified from the KPNC Diabetes Registry in the study 1.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Full Cohort
Number analyzed (Participants) | 236507
Ratio
  Prostate: 1-9000 mg | 1.08 [0.91 to 1.27]
  Prostate: 9001-25000 mg | 1.24 [1.06 to 1.46]
  Prostate: 25001-50000 mg | 1.12 [0.92 to 1.37]
  Prostate: >=50001 mg | 1.00 [0.78 to 1.28]
  Breast: 1-9000 mg | 0.89 [0.73 to 1.08]
  Breast: 9001-25000 mg | 0.95 [0.77 to 1.17]
  Breast: 25001-50000 mg | 1.15 [0.91 to 1.46]
  Breast: >=50001 mg | 1.19 [0.89 to 1.57]
  Lung/Bronchus: 1-9000 mg | 0.98 [0.80 to 1.21]
  Lung/Bronchus: 9001-25000 mg | 0.91 [0.73 to 1.15]
  Lung/Bronchus: 25001-50000 mg | 0.97 [0.75 to 1.26]
  Lung/Bronchus: >=50001 mg | 1.12 [0.84 to 1.50]
  Colon: 1-9000 mg | 0.87 [0.69 to 1.10]
  Colon: 9001-25000 mg | 0.86 [0.68 to 1.10]
  Colon: 25001-50000 mg | 0.97 [0.74 to 1.27]
  Colon: >=50001 mg | 0.79 [0.56 to 1.12]
  Non-Hodgkin Lymphoma: 1-9000 mg | 0.92 [0.66 to 1.29]
  Non-Hodgkin Lymphoma: 9001-25000 mg | 1.16 [0.85 to 1.59]
  Non-Hodgkin Lymphoma: 25001-50000 mg | 1.02 [0.69 to 1.51]
  Non-Hodgkin Lymphoma: >=50001 mg | 0.66 [0.38 to 1.13]
  Corpus Uteri: 1-9000 mg | 1.02 [0.76 to 1.37]
  Corpus Uteri: 9001-25000 mg | 0.90 [0.64 to 1.25]
  Corpus Uteri: 25001-50000 mg | 0.67 [0.42 to 1.06]
  Corpus Uteri: >=50001 mg | 0.87 [0.54 to 1.42]
  Pancreatic: 1-9000 mg | 1.50 [1.14 to 1.98]
  Pancreatic: 9001-25000 mg | 1.10 [0.79 to 1.53]
  Pancreatic: 25001-50000 mg | 1.46 [1.04 to 2.06]
  Pancreatic: >=50001 mg | 1.61 [1.10 to 2.35]
  Kidney/Renal Pelvis: 1-9000 mg | 0.83 [0.57 to 1.19]
  Kidney/Renal Pelvis: 9001-25000 mg | 1.03 [0.73 to 1.44]
  Kidney/Renal Pelvis: 25001-50000 mg | 0.86 [0.56 to 1.32]
  Kidney/Renal Pelvis: >=50001 mg | 1.05 [0.67 to 1.64]
  Rectum: 1-9000 mg | 0.84 [0.54 to 1.30]
  Rectum: 9001-25000 mg | 0.76 [0.47 to 1.23]
  Rectum: 25001-50000 mg | 0.75 [0.42 to 1.34]
  Rectum: >=50001 mg | 0.82 [0.41 to 1.61]
  Melanoma: 1-9000 mg | 1.20 [0.84 to 1.72]
  Melanoma: 9001-25000 mg | 1.26 [0.88 to 1.81]
  Melanoma: 25001-50000 mg | 1.03 [0.66 to 1.62]
  Melanoma: >=50001 mg | 1.14 [0.70 to 1.85]

8. Secondary Outcome: Number of 10 Most Common Cancer Cases By Dose of Pioglitazone
Description: The 10 most common cancer cases included: prostate, female breast, lung/bronchus, endometrial, colon, non-Hodgkin lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma associated with dose of pioglitazone. The various doses include 1-9000 mg, 9001-25000 mg, 25001-50000 mg and >=50001 mg.
Time Frame: 15 years 5 months
Population: Analysis population included T2DM participants who were identified from the KPNC Diabetes Registry in the study 1.The unexposed arm was not planned to be analyzed for this outcome measure.
Measure: Number; unit: Cases
Arm/Group | Ever User of Pioglitazone
Number analyzed (Participants) | 38190
Cases
  Prostate: 1-9000 mg | 129
  Prostate: 9001-25000 mg | 167
  Prostate: 25001-50000 mg | 109
  Prostate: >=50001 mg | 71
  Breast: 1-9000 mg | 92
  Breast: 9001-25000 mg | 98
  Breast: 25001-50000 mg | 77
  Breast: >=50001 mg | 53
  Lung/Bronchus: 1-9000 mg | 90
  Lung/Bronchus: 9001-25000 mg | 81
  Lung/Bronchus: 25001-50000 mg | 61
  Lung/Bronchus: >=50001 mg | 50
  Colon: 1-9000 mg | 72
  Colon: 9001-25000 mg | 70
  Colon: 25001-50000 mg | 56
  Colon: >=50001 mg | 35
  Non-Hodgkin Lymphoma: 1-9000 mg | 34
  Non-Hodgkin Lymphoma: 9001-25000 mg | 44
  Non-Hodgkin Lymphoma: 25001-50000 mg | 28
  Non-Hodgkin Lymphoma: >=50001 mg | 14
  Corpus Uteri: 1-9000 mg | 43
  Corpus Uteri: 9001-25000 mg | 38
  Corpus Uteri: 25001-50000 mg | 19
  Corpus Uteri: >=50001 mg | 18
  Pancreatic: 1-9000 mg | 52
  Pancreatic: 9001-25000 mg | 39
  Pancreatic: 25001-50000 mg | 38
  Pancreatic: >=50001 mg | 32
  Kidney/Renal Pelvis: 1-9000 mg | 28
  Kidney/Renal Pelvis: 9001-25000 mg | 37
  Kidney/Renal Pelvis: 25001-50000 mg | 23
  Kidney/Renal Pelvis: >=50001 mg | 22
  Rectum: 1-9000 mg | 20
  Rectum: 9001-25000 mg | 18
  Rectum: 25001-50000 mg | 12
  Rectum: >=50001 mg | 9
  Melanoma: 1-9000 mg | 28
  Melanoma: 9001-25000 mg | 34
  Melanoma: 25001-50000 mg | 21
  Melanoma: >=50001 mg | 19

ADVERSE EVENTS:
Description: Due to the observational nature of study individual adverse events (AEs) were not planned to be collected and reported.
Arm/Group | Ever User of Pioglitazone | Never User of Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.